CLINICAL TRIAL: NCT03264534
Title: Manually Performed Limbal Relaxing Incisions vs Femtosecond Laser-guided Astigmatic Keratotomy for Correction of Corneal Astigmatism After Phacoemulsification
Brief Title: Manually Performed Limbal Relaxing Incisions vs Femtosecond Laser-guided Astigmatic Keratotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ashraf Rashwan, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17200119
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Corneal Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- limbal relaxing incisions (Active Comparator): Manually performed limbal relaxing incisions
  Interventions: Procedure: limbal relaxing incisions
- astigmatic keratotomy (Active Comparator): femtosecond laser-guided astigmatic keratotomy
  Interventions: Procedure: astigmatic keratotomy

INTERVENTIONS:
Procedure: limbal relaxing incisions — Manually performed surgical procedure
  Arms: limbal relaxing incisions
Procedure: astigmatic keratotomy — femtosecond laser guided surgical procedure
  Arms: astigmatic keratotomy

SUMMARY:
Astigmatic keratotomy (AK) is used to treat numerous refractive disorders, including congenital astigmatism, residual corneal astigmatism at the time of or following cataract surgery, post-traumatic astigmatism, and astigmatism after corneal transplantation.

Within the past few years, much consideration has been given to an evolutionary variant of the procedure, the limbal relaxing incision (LRI). By moving the incision farther to the periphery, cataract surgeons can safely and predictably remediate mild to moderate amounts of regular astigmatism at the time of cataract surgery by performing this incisional technique.

Recent technological developments have shifted ophthalmologist's attention from manually created LRIs and astigmatic keratotomy procedures to femtosecond laser-guided procedures. Femtosecond lasers offer superior incisional accuracy and reproducibility coupled with minimal effects on collateral tissues, achieving levels of safety and reproducibility exceeding those of mechanical techniques. A major clinical application of the femtosecond laser is for creating arcuate incisions that have a precise and accurate length, depth, angular position, and optical zone.

DETAILED DESCRIPTION:
Pre-operative evaluation:

1. Close examination of the peripheral cornea by slit lamb, particularly in the areas where the incisions will be placed.
2. Fundus examination to exclude other causes of diminution of vision.
3. IOP measure.
4. Precise manifest refraction, uncorrected visual acuity and best corrected visual acuity by snellen's chart.
5. Standard keratometry to confirm diopters of corneal astigmatism.
6. Corneal Tomography (Pentacam).

Surgical procedures:

LRIs are performed using topical anesthesia. Patients are instructed to fixate on the microscope light. Before surgery, the steep meridian was identified with a marker dyed with methylene blue with the patient sitting up right. A diamond knife is set at a depth of 0.600 mm to 0.650 mm based on the peripheral pachymetric readings over the area of intended incision. The goal was a maximum reduction in astigmatism without overcorrection in with-the rule cases and with little overcorrection in against the rule cases. In the case of an overcorrection, the LRI can be sutured without creating any irregular astigmatism.

Performing femtosecond laser-guided astigmatic keratotomy requires the parameters of length, position, depth and distance from the visual axis where the incisions will be created. The depth of our incisions is 85% of the corneal pachymetry in the area of the incision. We have set our distance from the visual axis at 8 mm. This information is all downloaded onto the femtosecond laser. Then, we begin the surgical procedure by docking the laser onto the cornea. An overlay of the incisions is then visible on the surgical screen. After treatment, we bring the patient to the operating microscope and open the incisions with a Sinskey hook. By using low energy, the incisions do not have significant effect until they are opened.

ELIGIBILITY:
Inclusion Criteria:

1. patients who have undergo phacoemulsification.
2. Clear cornea.
3. Astigmatism from 1 diopter up to 4 diopters

Exclusion Criteria:

1. corneal opacity.
2. History of corneal surgery.
3. Thin cornea.
4. Other cause of diminution of vision rather than corneal astigmatism (eg: optic disc atrophy & maculopathy).
5. Astigmatism less than 1 diopter and more than 4 diopters.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Keratometric reading | 1 week
  measured by Corneal Tomography (Pentacam)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
There is a possibility of using these data in another related study so i am not sure about the time of sharing the individual participant data